CLINICAL TRIAL: NCT03965481
Title: Comparing Accuracy of PET/MR vs. CECT in Assessment of Peritoneal Disease for Resectability in Patients With Ovarian Cancer or Highly Suspected Ovarian Cancer
Brief Title: PET/MR Versus CECT Scans in Imaging Patients With Ovarian Cancer or Highly Suspected Ovarian Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017-0442; NCI-2019-02455 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-0442 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-05-24; First posted 2019-05-29 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Malignant Ovarian Neoplasm; Ovarian Carcinoma
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic (CECT, PET-MRI) (Experimental): Patients undergo standard of care CECT scan and PET-MRI scan over 90-120 minutes within 30 days before laparoscopy or cytoreduction. Patients who do not undergo cytoreduction based on diagnostic laparoscopy undergo additional PET-MRI and standard of care CECT scans after completion of chemotherapy and before cytoreduction.
  Interventions: Radiation: Dynamic Enhanced CT; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography

INTERVENTIONS:
Radiation: Dynamic Enhanced CT — Undergo standard CECT
  Other Names: Contrast-Enhanced Spiral CT; Dynamic Contrast Enhanced Computed Tomography; Dynamic Contrast Enhanced CT; Dynamic Contrast Material Enhanced CT; Dynamic Enhanced Computed Tomography; Enhanced Spiral CT
Procedure: Magnetic Resonance Imaging — Undergo PET/MRI scan
  Other Names: Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging
Procedure: Positron Emission Tomography — Undergo PET/MRI scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging

SUMMARY:
This trial studies how well positron emission tomography/magnetic resonance (PET/MR) versus contrast enhanced computerized tomography (CECT) scans work in locating ovarian cancer tumors in patients with known or suspected ovarian cancer. PET, MR, and CECT scans use different methods to create images of areas inside the body. This trial is being done to see if PET/MR scans may help doctors locate ovarian cancer tumors, predict how well these tumors may be removed during surgery, and predict how patients respond to platinum-based chemotherapies compared to standard of care CECT scans.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare PET/MR and contrast enhanced computed tomography (CT) to determine the accuracy in patients with advanced-stage serous ovarian cancer or highly suspected ovarian cancer using diagnostic laparoscopy as the gold standard with respect to lesion detection.

SECONDARY OBJECTIVES (EXPLORATORY):

I. Correlating imaging findings such as enhancement pattern, apparent diffusion coefficient (ADC) values, standardized uptake value (SUV) values, and advanced image analytics such as texture with pathology and genomic analysis for those lesions evaluated as a discovery arm.

II. Assess whether MR (multiparametric and functional) and PET findings predict response to platinum based chemotherapy.

III. To compare PET/MR and contrast enhanced CT to predict tumor negative (R0) resection using surgery as the gold standard.

OUTLINE:

Patients undergo standard of care CECT scan and PET-MRI scan over 90-120 minutes within 30 days before laparoscopy or cytoreduction. Patients who do not undergo cytoreduction based on diagnostic laparoscopy undergo additional PET-MRI and standard of care CECT scans after completion of chemotherapy and before cytoreduction.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ovarian cancer or highly suspected ovarian cancer who are eligible to undergo laparoscopic evaluation for resectability will be enrolled in the trial.
* Patients who have estimated glomerular filtration rate (eGFR) > 30.

Exclusion Criteria:

* Patients allergic to gadolinium.
* Patients who have eGRF < 30.
* Patients with cardiac pacers.
* Pediatric patients.
* Greater than 400 pounds in weight.
* Blood glucose (> 200 mg/dl).
* Pregnant women.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-05-12 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Lesion detection accuracy | Up to 3 years
  Lesion detection accuracy will be summarized using frequencies and percentages by modality. McNemar's test will be used to compare accuracies between positron emission tomography (PET)/magnetic resonance (MR) and contrast enhanced computerized tomography (CECT). Other diagnostic metrics (sensitivity, specificity, positive predictive value, and negative predictive value) will be estimated along with 95% confidence intervals. Logistic regression model will be used to assess effect of patient and tumor characteristics on diagnostic accuracy.

SECONDARY OUTCOMES:
Diagnostic accuracy by location | Up to 3 years
  Will be analyzed using linear regression or generalized linear regression models where applicable.
Response status | Up to 3 years
  Will be analyzed using linear regression or generalized linear regression models where applicable.
Imaging and genomic data analysis | Up to 3 years
  Correlation between imaging and genomic data will be analyzed using linear regression or generalized linear regression models where applicable.

CONTACTS AND LOCATIONS:
Overall Officials: Priya R Bhosale, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org